CLINICAL TRIAL: NCT05376527
Title: Open Multi-cohort Study of the First Phase of Safety of a Drug Based on Double Recombinant Vaccinia Virus VV-GMCSF-Lact in Patients With Recurrent/Refractory Metastatic Breast Cancer With Single and Multiple Administration
Brief Title: Open Multi-cohort Study of the First Phase of Safety of a Drug Based on Double Recombinant Vaccinia Virus VV-GMCSF-Lact
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: "Oncostar" LLC (Industry)
Collaborators: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Oncolact2020
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Oncolytic Virotherapy
Keywords: vaccinia virus; breast cancer; GMCSF; Lactaptin
MeSH Terms: conditions — Vaccinia; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Open Multi-cohort Study of Safety and Tolerability
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VV-GMCSF-Lact (Experimental): Double Recombinant Vaccinia Virus VV-GMCSF-Lact
  Interventions: Biological: Double Recombinant Vaccinia Virus VV-GMCSF-Lact

INTERVENTIONS:
Biological: Double Recombinant Vaccinia Virus VV-GMCSF-Lact — Intratumoral injections:
  1*107 PFU (calculated at minimal ED on mice); 2*107 PFU; 4*107 PFU; 6*107 PFU; 8*107 PFU; 10*107 PFU;

SUMMARY:
Purpose of the study is to evaluate the safety, tolerability and pharmacokinetic parameters of the drug based on double recombinant vaccinia virus VV-GMCSF-Lact, in patients with recurrent/refractory metastatic breast cancer in successive cohorts with dose escalation with single and multiple administration.

The study provides: determination of the maximum tolerated dose of the drug and the frequency, nature, intensity and duration of adverse events connected with the use of the study drug in escalating doses; detection of dose-limiting toxicity, its severity, duration and reversibility; determination of the profile of virus pharmacokinetics and antivirus antibodies; assessment of the objective response to the treatment.

Stage 1,: The virus drug is administered intratumorally once according to a "3+3" design in the dosage from 1*107 PFU to 10*107 PFU. The frequency of dose-limiting toxicity (DLT) will be evaluated (non-hematological toxicity III degree and above; development of febrile neutropenia and body temperature > 38.3°C more than two days after drug administration; thrombocytopenia III degree and above and/or hemorrhagic complications; repeated increase in ALT and/or AST activity is more than 4 times higher than the normal upper limit).

Escalation to the next level occurs if there is no DLT in the entire cohort under study. The study stops if the incidence of DLT in a cohort of 3 patients is 2 or 3. The maximum tolerated dose (MTD) will be considered the studied dose that is lower than the dose which DLT was determined. Stage 1 assumes randomization of no more than 36 patients.

Stage 2, multiple administration: According to Stage 1 the study will move to the second stage if there will be possibility to study at least one dosage regimen based on the previously studied dose. At Stage 2 two doses in ascending order below the MTD and MTD are planned to be used. Escalation to the next level occurs if no DLT is observed during dosing of the first three patients. If DLT develops and drug administration is discontinued, the patient is not excluded from the study, her drug administration visits are skipped, and she goes through all follow-up visits. The drug will be administered intratumorally 1 time per week for 4 weeks in 3 dosages: MTD and 2 lower dosages. Each cohort will include up to 6 patients in a "3+3" design. It is expected to include up to 24 patients, taking into account the possible inclusion of patients to replace those who left.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with recurrent and/or metastatic breast cancer, for whom the standard methods of treatment are considered ineffective by the medical commission.
2. Histologically confirmed progressive / metastatic tumor.
3. Detectable and measurable tumor foci - at least one measurable tumor site measured by CT (with a diameter more than 1 cm) and at least one tumor site for biopsy.
4. Body weight index from 18.5 to 30 kg / m2 with body weight from 55 to 100 kg inclusive.
5. Before inclusion of patients in the study, at least one of the following types of therapy was previously performed:

   5.1 previous radiation therapy completed more than 4 weeks ago before the screening visit; 5.2 previous immunotherapy completed more than 4 weeks ago before the screening visit; 5.3 previous hormone therapy completed more than 4 weeks ago before the screening visit; 5.4 previous chemotherapy completed more than 4 months ago before the screening visit.
6. The indicator of general status is not more than 2 points according the WHO scale.
7. Age - 18 years or older.
8. The level of ALT and AST does not exceed the upper limits of normal values more than 4 times.
9. Hematological parameters: the number of leukocytes > 3000/µl, platelets > 100000/µl, hemoglobin > 8 g/DL.
10. Negative result of the PCR test for the presence of SARS-CoV-2 virus RNA on screening.
11. No signs of SARS at least 14 days before screening.
12. Patients, 12.1. Not vaccinated against the SARS-CoV-2 coronavirus. OR 12.2. Vaccinated/revaccinated against SARS-CoV-2 coronavirus more than 90 days before the screening visit.
13. Patient's ability to perform the study procedure and provide written informed consent in accordance with the GCP and local laws.

Exclusion Criteria:

1. Incompatibility of patients with the inclusion criteria mentioned above.
2. Severe cardiovascular diseases in the past and at the present time (myocardial infarction, hypertension, stroke, phlebothrombosis, coronary insufficiency requiring medical correction, etc.).
3. Allergic reactions to any pharmacological drugs.
4. Positive reaction of serological study to HIV, hepatitis B and C, syphilis.
5. The use of immunosuppressive therapy for 90 days before inclusion in the study.
6. Myeloproliferative disorders requiring systemic therapy, according to anamnesis.
7. Exfoliative skin diseases (e.g. eczema or atopic dermatitis) requiring systemic therapy, according to anamnesis.
8. Clinically significant renal pathology (bilateral renal artery stenosis, renal artery stenosis in a single kidney, patients undergoing kidney transplantation, clinically significant decrease in sodium, hypo- or hyperglycemia, creatinine exceeding the upper limit of normal values more than 2 times).
9. Impaired renal function (decreased glomerular filtration rate less than 40 ml / min / 1,73 m2, estimated by the CKD-EPI calculation method).
10. Absence of adequate venous access, allowing to perform infusion therapy.
11. The inability of the CT.
12. Use of drugs or therapies listed in the Prohibited Therapies section.
13. The need for any vaccination/revaccination during the study.
14. Mental illness that prevents the patient from understanding the treatment plan.
15. Persons with alcohol, drug or drug addiction
16. Pregnancy or breastfeeding, refusal of a reliable method of contraception.
17. The need to use therapy during the study that is not permitted by this protocol.
18. Any clinical condition or deviation from normal laboratory and vital signs at screening that, in the opinion of the Investigator, would preclude the safe completion of the study protocol.
19. Participation in other clinical trials currently or within the last 3 months.
20. Previous serious systemic reaction or adverse effect from a previous smallpox vaccination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Frequency, nature, intensity and duration of adverse events related with the use of the study drug | 90 days from the data of the last treatment (for Stage 1 up to 107 days from participation in the study; for Stage 2 up to 129 days from participation in the study
  The severity of adverse events will be assessed according to CTCAE (Common Terminology Criteria for Adverse Events) Version 5.0. National Cancer Institute. 2017.
Degree of severity, duration, reversibility of dose-limiting toxicity | plus 3 days to the day of the last treatment
  Degree of severity, duration and reversibility of dose-limiting toxicity will be detected

SECONDARY OUTCOMES:
Determination of virus concentrations in blood | up to 216 hours to the last treatment
  Determination of virus concentrations in blood after 5, 15, 30 minutes, 1, 3, 6, 12, 24, 48, 72, 120, 168 and 216 hours after intratumoral administration

OTHER OUTCOMES:
Determination of the antivirus antibodies titer in the blood | up to 28 days to the last treatment
  Determination of the antivirus antibodies titer in the blood after 7, 14, 21, 28 days after intratumoral administration.
Assessment of Objective response (stabilization / progression rate) to treatment. Evaluation of tumor size | up to 107 days from participation in the study for Stage 1; up to 129 days from participation in the study for Stage 2
  Assessment of Objective response (stabilization / progression rate) to treatment on the RECIST 1.1 scale.
  Evaluation of tumor size according to the results of CT.

CONTACTS AND LOCATIONS:
Overall Officials: Petr V. Krivorotko, Professor, Principal Investigator — N.N. Petrov National Medical Research Center of Oncology
Locations (1):
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia